CLINICAL TRIAL: NCT01793831
Title: Efficacy and Safety of Standardized Fecal Microbiota Transplantation for Moderate to Severe Crohn's Diseases
Brief Title: Standardized Fecal Microbiota Transplantation for Crohn's Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Collaborators: The Affiliated Huaian NO.1 People's Hospital of Nanjing Medical University (Unknown); The First Affiliated Hospital of Air Force Medicial University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Associate professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMC-CN-121101
Record Dates: First submitted 2013-02-13; First posted 2013-02-18 (Estimated); Last update posted 2024-11-29 (Actual); Status verified 2024-08

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease (CD)
Keywords: Inflammatory bowel disease; Fecal transplantation; Fecal bacteriotherapy; Fecal microbiota transplantation; Crohn's disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fecal microbiota transplantation (Experimental): Standard fecal microbiota transplantation, which has been defined as washed microbiota transplantation since 2019.
  Interventions: Procedure: FMT
- Traditional treatments (No Intervention): Traditional treatments for Crohn's disease and its complications according to the guidelines.

INTERVENTIONS:
Procedure: FMT — Standard FMT
  Arms: Fecal microbiota transplantation

SUMMARY:
The gut microbiota is considered to constitute a "microbial organ" which has pivotal roles in the intestinal diseases and body's metabolism. Evidence from animal and human studies strongly supports the link between intestinal bacteria and inflammatory bowel diseases (IBD). Dozens of studies reported its efficacy in treatment of severe Clostridium difficile colitis. Preliminary studies using fecal microbiota transplantation (FMT) for Ulcerative Colitis (UC), Crohn's diseases (CD), irritable bowel syndrome (IBS) and constipation have also met with some success. However, the results on CD is very limited. This marks the initial step in exploring the potential efficacy of fecal bacteriotherapy for CD. The investigators aim to evaluate the effectiveness, durability, and safety of FMT in a cohort of at least 500 patients with CD over a ten-year period

DETAILED DESCRIPTION:
The present clinical trial aims to re-establish a gut functionality state of intestinal flora through FMT as a therapy for CD (all age range,HBI>4). We established a standard microbiota isolation from donated fresh stool in lab. The microbiota is then transplanted into the intestine via endoscopy or other established methods, such as mid-gut or colonic transendoscopic enteral tubing. Patients from multi-clinical centers in this study will be assigned to receive FMT or traditional treatments according to associated guidelines and follow-up for at least one year. Blood tests, imaging, endoscopy and questionnaire will be used to assess participants at study start and at study completion.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Crohn's disease, with the diagnosis remaining unchanged after at least three months of follow-up.

Willingness to undergo FMT (Fecal Microbiota Transplantation).

Exclusion Criteria:

Presence of serious conditions that made them unsuitable for inclusion (e.g., malignant neoplasms, cardiopulmonary failure, serious liver or kidney disease).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinical remission | Up to one year
  Clinical remission defined as HBI score ≦ 4. For patients with complications such as intestinal obstruction, Clinical remission can be defined as obstruction improvement. The endpoint of follow-up is the time of clinical recurrence.

SECONDARY OUTCOMES:
Costs | Up to one year
  Social and medical costs
Adverse events | During FMT and ten years after FMT
  All possible adverse events:fever,abdominal pain,infectious diseases and others
Sleep quality | before FMT, 1 month after FMT, 12 weeks after FMT
  evaluated by Pittsburgh Sleep Quality Index (PSQI), with a score range of 0 to 21. Higher PSQI score indicates poorer sleep quality. Insomnia Severity Index (ISI), with a score range of 0 to 28. Higher ISI score indicates more severe insomnia.
Fatigue | before FMT, 1 month after FMT, 12 weeks after FMT
  evaluated by Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F), with a score range of 0 to 52. Higher FACIT-F score indicates lower levels of fatigue and better quality of life.
Anxiety and depression | before FMT, 1 month after FMT, 12 weeks after FMT
  evaluated by Hospital Anxiety and Depression Scale (HADS), with a score range of 0 to 42. Higher scores indicate greater severity of anxiety and depression symptoms.
Symptomatic stricture | before FMT, 1 month after FMT, 12 weeks after FMT
  evaluated by Crohn's Disease Obstruction Score (CDOS), with a score range of 0 to 6. Higher scores indicate greater severity of obstructive symptoms.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Affiliated Huaian No.1 People's Hospital of Nanjing Medical University, Huai'an, Jiangsu
  - Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu

REFERENCES:
- [Background] Damman CJ, Miller SI, Surawicz CM, Zisman TL. The microbiome and inflammatory bowel disease: is there a therapeutic role for fecal microbiota transplantation? Am J Gastroenterol. 2012 Oct;107(10):1452-9. doi: 10.1038/ajg.2012.93. PMID 23034604
- [Background] Aroniadis OC, Brandt LJ. Fecal microbiota transplantation: past, present and future. Curr Opin Gastroenterol. 2013 Jan;29(1):79-84. doi: 10.1097/MOG.0b013e32835a4b3e. PMID 23041678
- [Background] Zhang FM, Wang HG, Wang M, Cui BT, Fan ZN, Ji GZ. Fecal microbiota transplantation for severe enterocolonic fistulizing Crohn's disease. World J Gastroenterol. 2013 Nov 7;19(41):7213-6. doi: 10.3748/wjg.v19.i41.7213. PMID 24222969
- [Background] Zhang T, Xiang J, Cui B, He Z, Li P, Chen H, Xu L, Ji G, Nie Y, Wu K, Fan D, Huang G, Bai J, Zhang F. Cost-effectiveness analysis of fecal microbiota transplantation for inflammatory bowel disease. Oncotarget. 2017 Oct 4;8(51):88894-88903. doi: 10.18632/oncotarget.21491. eCollection 2017 Oct 24. PMID 29179485
- [Background] He Z, Li P, Zhu J, Cui B, Xu L, Xiang J, Zhang T, Long C, Huang G, Ji G, Nie Y, Wu K, Fan D, Zhang F. Multiple fresh fecal microbiota transplants induces and maintains clinical remission in Crohn's disease complicated with inflammatory mass. Sci Rep. 2017 Jul 6;7(1):4753. doi: 10.1038/s41598-017-04984-z. PMID 28684845
- [Background] Cui B, Feng Q, Wang H, Wang M, Peng Z, Li P, Huang G, Liu Z, Wu P, Fan Z, Ji G, Wang X, Wu K, Fan D, Zhang F. Fecal microbiota transplantation through mid-gut for refractory Crohn's disease: safety, feasibility, and efficacy trial results. J Gastroenterol Hepatol. 2015 Jan;30(1):51-8. doi: 10.1111/jgh.12727. PMID 25168749
- [Derived] Lu G, Zhang S, Wang R, Wu X, Chen Y, Wen Q, Cui B, Zhang F, Li P. Fecal microbiota transplantation improves bile acid malabsorption in patients with inflammatory bowel disease: results of microbiota and metabolites from two cohort studies. BMC Med. 2025 Sep 1;23(1):511. doi: 10.1186/s12916-025-04353-y. PMID 40890737
- [Derived] Li Q, Liu Y, Zhang Z, Zhang S, Ding X, Zhang F. Washed Microbiota Transplantation Improves the Sleep Quality in Patients with Inflammatory Bowel Disease. Nat Sci Sleep. 2024 Aug 2;16:1141-1152. doi: 10.2147/NSS.S460882. eCollection 2024. PMID 39109266
- [Derived] Li Q, Ding X, Liu Y, Marcella C, Dai M, Zhang T, Bai J, Xiang L, Wen Q, Cui B, Zhang F. Fecal Microbiota Transplantation is a Promising Switch Therapy for Patients with Prior Failure of Infliximab in Crohn's Disease. Front Pharmacol. 2021 May 17;12:658087. doi: 10.3389/fphar.2021.658087. eCollection 2021. PMID 34079458
- [Derived] Zhang T, Li P, Wu X, Lu G, Marcella C, Ji X, Ji G, Zhang F. Alterations of Akkermansia muciniphila in the inflammatory bowel disease patients with washed microbiota transplantation. Appl Microbiol Biotechnol. 2020 Dec;104(23):10203-10215. doi: 10.1007/s00253-020-10948-7. Epub 2020 Oct 16. PMID 33064186
- [Derived] Xiang L, Ding X, Li Q, Wu X, Dai M, Long C, He Z, Cui B, Zhang F. Efficacy of faecal microbiota transplantation in Crohn's disease: a new target treatment? Microb Biotechnol. 2020 May;13(3):760-769. doi: 10.1111/1751-7915.13536. Epub 2020 Jan 20. PMID 31958884
- [Derived] Li P, Zhang T, Xiao Y, Tian L, Cui B, Ji G, Liu YY, Zhang F. Timing for the second fecal microbiota transplantation to maintain the long-term benefit from the first treatment for Crohn's disease. Appl Microbiol Biotechnol. 2019 Jan;103(1):349-360. doi: 10.1007/s00253-018-9447-x. Epub 2018 Oct 24. PMID 30357440